CLINICAL TRIAL: NCT01295320
Title: Long Term Immunogenicity and Safety of GSK Biologicals' Herpes Zoster Vaccine 1437173A in Healthy Subjects
Brief Title: Study of Long Term Immune Responses and Safety of the GSK Herpes Zoster Vaccine in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 114825
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Results first posted 2017-10-05 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-10

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster; vaccine; safety; immunogenicity
MeSH Terms: conditions — Herpes Zoster | interventions — Blood Specimen Collection

ARMS (1):
- GSK1437173A Group (Experimental): Subjects who received 2 doses of HZ vaccine in the intermediate dose study group in study 108494 (NCT00434577). No treatment was given in this current study (NCT01295320).
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Blood sample will be collected at Month 48, Month 60 and Month 72

SUMMARY:
The subjects included in this study are subjects that participated in study NCT00434577. These subjects were vaccinated with the candidate Herpes Zoster (HZ) vaccine at Month 0 and Month 2 and were then followed at Month 12, Month 24 and Month 36 (study NCT00434577) for safety and immunogenicity.

This long term follow up study (ZOSTER-024 [114825]) will evaluate immune responses to and safety of the previously administered candidate HZ vaccine at Months 48, 60 and 72.

The study visits will be scheduled at approximately one year intervals after the first visit in ZOSTER-024. Blood samples for the evaluation of cellular and humoral immunity will be taken from all subjects at each visit. Information on safety and the occurrence of HZ will also be collected during these visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol
* Previous participation in study NCT00434577 as a member of the intermediate dose active vaccine group
* Written informed consent obtained from the subject

Exclusion Criteria:

* Having participated in another study at any time after NCT00434577 study end in which the subject was exposed to an investigational or non-investigational product or; concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first blood draw
* Having received a vaccine containing some vaccine components, any time after study end of study NCT00434577
* Having received a vaccine against HZ any time after study end of study NCT00434577
* Subject who did not receive a complete vaccination course of 2 doses of the intermediate dose active vaccine in study NCT00434577

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-02-28 (Actual); Primary Completion 2013-06-20 (Actual); Study Completion 2013-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- GSK Investigational Site, Hradec Králové, Czechia
- Germany (6):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Rotterdam
- Sweden (2):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK1437173A Group
Started | 129
Completed | 119
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2
Not completed — Subject was bedridden | 1
Not completed — Unable to travel | 1

BASELINE CHARACTERISTICS:
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.8 (4.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian/European Heritage | 128
  African Heritage/African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Cell-Mediated Immunity (CMI) in Terms of Frequencies of Antigen-specific CD4 T Cells
Description: -Frequencies of CD4 T cells with antigen-specific Interferon gamma (IFN-γ) and/or Interleukin-2 (IL-2) and/or Tumour Necrosis Factor alpha (TNF-α) and/or CD40 Ligand (CD40L) secretion/expression to glycoprotein E (gE) and Varicella Zoster Virus (VZV) as determined by Intracellular Cytokine Staining (ICS)
Time Frame: Month 48
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures defined in the protocol and with no elimination criteria during the study).
Measure: Mean (Standard Deviation); unit: cells/million T-cells
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 126
cells/million T-cells
  CD4[2+] anti-gE specific cells: number analyzed (Participants) | 118
  CD4[2+] anti-gE specific cells | 726.19 (1051.77)
  CD4[2+] anti-VZV specific cells: number analyzed (Participants) | 118
  CD4[2+] anti-VZV specific cells | 567.52 (531.31)

2. Primary Outcome: Cell-Mediated Immunity (CMI) in Terms of Frequencies of Antigen-specific CD4 T Cells
Description: Frequencies of CD4 T cells with antigen-specific Interferon gamma (IFN-γ) and/or Interleukin-2 (IL-2) and/or Tumour Necrosis Factor alpha (TNF-α) and/or CD40 Ligand (CD40L) secretion/expression to glycoprotein E (gE) and Varicella Zoster Virus (VZV) as determined by Intracellular Cytokine Staining (ICS)
Time Frame: Month 60
Population: The analysis was base don the ATP cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures defined in the protocol and with no elimination criteria during the study).
Measure: Mean (Standard Deviation); unit: cells/million T-cells
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 126
cells/million T-cells
  CD4[2+] anti-gE cells: number analyzed (Participants) | 48
  CD4[2+] anti-gE cells | 744.43 (810.14)
  CD4[2+] anti-VZV cells: number analyzed (Participants) | 95
  CD4[2+] anti-VZV cells | 697.75 (550.17)

3. Primary Outcome: Cell-Mediated Immunity (CMI) in Terms of Frequencies of Antigen-specific CD4 T Cells
Description: as for outcome 2
Time Frame: Month 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/million T-cells
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 126
cells/million T-cells
  CD4[2+] anti-gE cells: number analyzed (Participants) | 75
  CD4[2+] anti-gE cells | 630.76 (548.14)
  CD4[2+] anti-VZV cells: number analyzed (Participants) | 76
  CD4[2+] anti-VZV cells | 473.06 (449.71)

4. Primary Outcome: Antigen-specific Antibody (Ab) Concentrations
Description: -Anti-Glicoprotein E (Anti-gE) and anti-VZV Ab concentrations as determined by Enzyme-Linked Immunosorbent Assay (ELISA)
Time Frame: Month 48
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 126
mIU/ml
  anti-gE | 9093.2 [8041.3 to 10282.6]
  anti-VZV: number analyzed (Participants) | 108
  anti-VZV | 2869.9 [2565.5 to 3210.5]

5. Primary Outcome: Antigen-specific Antibody (Ab) Concentrations
Description: as for outcome 4
Time Frame: Month 60
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 126
mIU/ml
  anti-gE: number analyzed (Participants) | 121
  anti-gE | 8831.3 [7767.2 to 10041.3]
  anti-VZV: number analyzed (Participants) | 95
  anti-VZV | 2890.0 [2536.0 to 3293.4]

6. Primary Outcome: Antigen-specific Antibody (Ab) Concentrations
Description: as for outcome 4
Time Frame: Month 72
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 126
mIU/ml
  anti-gE | 7711.3 [6810.8 to 8730.9]
  anti-VZV: number analyzed (Participants) | 107
  anti-VZV | 2933.4 [2577.7 to 3338.1]

7. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) Related to the Study Participation
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Month 48 to Month 72
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 129
Participants | 2

8. Secondary Outcome: Number of Subjects With Any SAEs Related to Previous Vaccination and Not Already Documented
Description: as for outcome 7
Time Frame: Month 0 to Month 72
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 129
Participants | 0

9. Secondary Outcome: Number of Subjects With Any Fatal SAEs
Description: as for outcome 7
Time Frame: Month 48 to Month 72
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 129
Participants | 2

10. Secondary Outcome: Number of Subjects With Any Suspected Cases of HZ Episodes
Time Frame: Month 48 to Month 72
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 129
Participants | 1

11. Secondary Outcome: Number of Subjects With Any Suspected Cases of HZ Episodes Following Participation in 108494 Study and Its Follow-ups (108516, 108518 and 108520) and Not Already Documented
Time Frame: Month 48 to Month 72
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 129
Participants | 0

12. Secondary Outcome: Number of Subjects and Relationship to Vaccination of Any Potential Immune Mediated Diseases (pIMDs) Following Participation in 108494 Study and Its Follow-ups (108516, 108518 and 108520) and Not Already Documented
Time Frame: Month 48 to Month 72
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 129
Participants
  Any pIMDs | 1
  Related pIMDs | 0

ADVERSE EVENTS:
Time Frame: SAEs: Month 0 to Month 72
Description: No Frequent Adverse events were collected during this study.
Arm/Group | GSK1437173A Group
All-Cause Mortality (participants affected / at risk) | 2/129
Serious Adverse Events (participants affected / at risk) | 4/129
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1437173A Group (N=129)
Anaemia (Blood and lymphatic system disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Death (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.